CLINICAL TRIAL: NCT01697436
Title: A Bioequivalence Study of Ribavirin Oral Solution (RO0209963) Versus the Reference Ribavirin Tablets (Copegus) Following Oral Administration in Healthy Adult Subjects
Brief Title: A Bioequivalence Study of an Oral Solution of Copegus (Ribavirin) Compared to Copegus Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BP28307
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Ribavirin

ARMS (4):
- Crossover Period 1 (Experimental)
  Interventions: Drug: ribavirin [Copegus]
- Crossover Period 2 (Experimental)
  Interventions: Drug: ribavirin [Copegus]
- Crossover Period 3 (Experimental)
  Interventions: Drug: ribavirin [Copegus]
- Crossover Period 4 (Experimental)
  Interventions: Drug: ribavirin [Copegus]

INTERVENTIONS:
Drug: ribavirin [Copegus] — tablet under fed condition
  Arms: Crossover Period 1
Drug: ribavirin [Copegus] — tablet under fasted condition
  Arms: Crossover Period 2
Drug: ribavirin [Copegus] — oral solution under fed condition
  Arms: Crossover Period 3
Drug: ribavirin [Copegus] — oral solution under fasted condition
  Arms: Crossover Period 4

SUMMARY:
This four-period, single-center, open-label, single-dose, randomized, cross-over study will assess the bioequivalence and safety of an oral solution of Copegus (ribavirin) compared to a Copegus tablet in healthy adult volunteers. Volunteers will be randomized to one of four sequences in which they will receive the treatment under fed and under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteers
* Able to participate and willing to give informed consent and comply with the study restrictions.
* Negative urine pregnancy test (for women of childbearing potential) documented at screening and within the 24-hour period prior to each dose of test drug
* All male subjects with female partners of childbearing potential must agree to use two reliable forms of contraception, one of which must be a physical barrier method, during the study and for 6 months thereafter
* Female subjects must be postmenopausal or surgically sterile or they must agree to use two reliable forms of contraception one of which must be a physical barrier method, during treatment and for 6 months thereafter
* Body mass index (BMI) <30 kg/m2

Exclusion Criteria:

* Pregnant or lactating women and male partners of females who are pregnant or lactating
* Positive test for drugs of abuse at screening and within the 24-hour period prior to each dose of test drug.
* History (within 3 months of screening) of alcohol consumption exceeding 2 standard units per day on average (1 standard unit = 10 grams of alcohol). Alcohol consumption will be prohibited at least 48 hours before screening and from at least 48 hours before Day -1 through the end of the study
* Confirmed systolic blood pressure (SBP) > 140 or < 90 mm Hg, and diastolic blood pressure (DBP) > 90 or < 50 mm Hg
* Resting pulse rate > 90 or < 45 beats per minute
* History or symptoms of any significant disease including (but not limited to) hematological, neurological, psychiatric, cardiovascular, respiratory, gastrointestinal, hepatic, or renal disorder
* History of active malignancy within the last 5 years, with the exception of localized or in situ carcinoma of the skin (e.g., skin basal or squamous cell carcinoma)
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at screening
* Use of any medications (prescription or over-the-counter, vitamin, mineral, herbal, and dietary supplements within 7 days, or less than 5 half-lives (whichever is longer) prior to randomization. Exceptions are acetaminophen (up to 2 g/day), ibuprofen (up to 1 g/day), and hormonal contraceptives.
* Clinically significant abnormalities in laboratory test results
* Participation in an investigational drug study within 60 days or in an investigational device study within 30 days prior to screening
* Donation of blood over 500 mL from 3 months prior to screening until the end of the study; donation of plasma from 7 days prior to screening until the end of the study
* Concomitant disease or condition that could interfere with, or for which the treatment of might interfere with, the conduct of the study or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this study
* Smoker of more than 10 cigarettes per day prior to screening or use of tobacco products equivalent to more than 10 cigarettes per day
* Clinically significant abnormalities in the pre-dose resting electrocardiograms
* Any confirmed significant allergic reactions against RBV or known or potential allergy or hypersensitivity to the non-active ingredients of the study drugs (non-active hay fever is acceptable)
* Individuals receiving ribavirin therapy within 6 months prior to study initiation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: area under the plasma concentration time curve | Periods 1-4: Predose and up to 192 hours post-dose
Pharmacokinetics: maximum plasma concentration | Periods 1-4: Predose and up to 192 hours post-dose

SECONDARY OUTCOMES:
Safety: incidence of adverse events | Approximately 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Lenexa, Kansas, United States